CLINICAL TRIAL: NCT03823027
Title: Open-label, Single-arm, Multicenter Study Investigating Performance and Safety of SiPore15™ in Obese and Overweight Subjects With Prediabetes or Newly Diagnosed Type 2 Diabetes
Brief Title: STAR Study Investigating Performance and Safety of the Medical Device SiPore15™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sigrid Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR01
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: PreDiabetes; Pre Diabetes; Prediabetic State; Type2 Diabetes; Type2 Diabetes Mellitus; Overweight; Obese
Keywords: Medical Device; Prediabetes; Type2 Diabetes; Silica; Metabolic risk factors
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The single-arm study is designed to collect data on changes over time, i.e. comparing the pre-treatment/baseline value with the value achieved after full treatment (12 weeks). Thus, each individual act as his/her own control. The study design has been discussed with notified bodies, and deemed appropriate as there is no state-of-the-art pharmacotherapy for treatment of prediabetes to compare with.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-arm (Experimental): The device will be taken before three daily main meals togteher with water. The dose will be escalated from 1g per main meal to the full dose of 3g per main meal. The device is provided in foil stick-packs packed in boxes with weekly supply. The treatment is for 12 weeks.
  Interventions: Device: SiPore15™

INTERVENTIONS:
Device: SiPore15™ — SiPore15™ is a taste- and odourless white powder, consisting of precisely engineered micrometre sized synthetic amorphous silicon dioxide. The device is made of pure silicon dioxide, SiO2, which has the CAS Number: 112926-00-8 and EC List number: 601-214-2.

SUMMARY:
The primary objective of STAR01 is to evaluate the performance and safety of the medical device (class IIb) SiPore15™ after a 12-week long treatment in the target population of obese and overweight subjects with prediabetes or newly diagnosed type 2 diabetes. The expected performance and safety of the device is based on the safety and efficacy results seen in an earlier First-in-Man (FIM) study. The safety and tolerability of SiPore15™ is based on the well-established and extensive use of food grade silicon dioxide and favorable data from the FIM study. Data on side-effects will be collected for verification of device safety. The study duration is 24 weeks in total, 12 weeks from baseline on investigational medicinal device (IMD) treatment, with additional 12 weeks off treatment. The study population is planned for forty (40) subjects to be enrolled, male and females, age >18 years and fulfilling all inclusion criteria but none of the exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Male or female aged ≥18 years on the day of screening.
3. Female subjects of childbearing potential must be on non-oral contraceptives, postmenopausal or sterile.
4. Prediabetes or newly diagnosed T2D (not on blood sugar lowering drugs) defined as HbA1c levels: ≥42 to ≤57 mmol/mol (≥6.0 to ≤7.5%-according to DCCT).
5. Body mass index (BMI) >25 kg/m2 and > or = 40 kg/m2.
6. Stable weight for 3 months (+/-5 kg).
7. No extreme changes in diet for the last 6 months such as anorexia, bulimia, etc.
8. Subject must be able and willing to attend all scheduled visits and comply with all study procedures with no planned holiday longer than 2 weeks during the 12 weeks of treatment.

Exclusion Criteria:

1. Diagnosed with type1 diabetes/Latent Autoimmune Diabetes in Adult (LADA) or secondary diabetes, as part of medical history or confirmed by laboratory test.
2. Previous or current Metformin treatment or other glucose reducing drug therapy within 3 months before screening visit.
3. Previous or current statin treatment or other blood lipid (LDL) reducing drug therapy, within 12 months before screening visit.
4. Previous or current medication known to cause weight loss or weight gain, such as systemic corticosteroids, thyroid hormones or Estrogen, within 1 month before screening visit.
5. Subjects who stopped smoking within 6 months before screening visit.
6. Diagnosed with chronic somatic diseases, except for obesity and treatment naive T2D, that in the opinion of the investigator may therefore affect metabolic and /or intestinal function (e.g. inflammatory bowel disease, intestinal dysfunction, pancreatic dysfunction, other causes of malabsorption, recent (past 6 months) neoplastic disease.
7. Any history of myocardial infarction or stroke within the 6 months before screening visit.
8. Anemia, donated blood or other major blood loss within 3 months from screening visit that in the opinion of the clinician may interfere with the study.
9. Pregnancy or breast feeding.
10. Allergies to silicon dioxide.
11. A diagnosed state that requires use of vitamin and/or mineral supplements during the study.
12. Previous major gastric surgery that may affect the study outcome, such as bariatric surgery.
13. Ongoing or unstable kidney condition with moderate to great reduction in glomerular filtration rate < 90 ml/min (GFR) that may affect metabolic parameters during the trial.
14. Ongoing or unstable liver condition that may cause changes in liver enzymes exceeding 2x upper normal levels.
15. Psychiatric or cognitive disorder and/or behavioral problems which in the opinion of the clinician may interfere with the study.
16. History of or ongoing alcohol or drug addiction.
17. Participation in any study involving an investigational drug or medical device within the past 30 days before the screening visit.
18. Belongs to a vulnerable population or has any condition such that his/her ability to provide informed consent, comply with the follow-up requirements, or provide self- assessments is compromised (e.g. homeless, developmentally disabled and prisoner).
19. Is a relative of the Investigator or an employee at the clinical study site.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Performance measured as changes in HbA1c | From week 1 to week 12
  To measure change in long-term blood glucose levels, HbA1c, from baseline (week 1) to end- -of-treatment (week 12).
Tolerability measured as evaluation of Adverse Events | From week 1 to week 14
  To assess safety and tolerability by evaluating the frequency and incidence of both adverse events (AEs) and device related adverse events (ADEs) during the study treatment and follow-up, from baseline (week 1) until week 14.

SECONDARY OUTCOMES:
Performance measured as changes in LDL-C | From week 1 to week 12
  To measure change in LDL-C blood levels from baseline (week 1) to week 6 and end-of- treatment (week 12).
Performance measured as changes in body fat % | From week 1 to week 12
  To measure change in body fat levels (bio electric impedance, BIA) from baseline (week 1) to week 6 and end-of-treatment (week 12).

OTHER OUTCOMES:
Exploratory Endpoint on Medical Device Usability | From week 1 to week 12
  To assess Medical Device Usability by collecting data:
  a. Collect information on Ease of use (Easy, neither/nor, difficult) at visit week 2, 6 and end-of -treatment.
Explorative Endpoint on changes in Cholesterol | From week 1 to week 12
  To measure change in total Cholesterol levels from baseline to week 6 and end-of-treatment.
Explorative Endpoint on changes in microbiome diversity (species not defined) | From week 1 to week 24
  To explore changes in microbiome by feces sampling for research at baseline and at week 24.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsi Pietiläinen, Prof., Study Chair — Gyllenberg Professor in Clinical Metabolism Obesity Research Unit University of Helsinki
Locations (2):
- Pihlajalinna Ite, Satucon OY, Kuopio, Finland
- Clinical Trial Consultants, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baek J, Robert-Nicoud G, Herrera Hidalgo C, Borg ML, Iqbal MN, Berlin R, Lindgren M, Waara E, Udden A, Pietilainen K, Bengtsson T. Engineered mesoporous silica reduces long-term blood glucose, HbA1c, and improves metabolic parameters in prediabetics. Nanomedicine (Lond). 2022 Jan;17(1):9-22. doi: 10.2217/nnm-2021-0235. Epub 2021 Dec 2. PMID 34854740
- See also: Information about the site and study in Kuopio, Finland — https://www.laaketutkimukseen.fi
- See also: Information about the site and study in Uppsala, Sweden — http://www.forskningsperson.se